CLINICAL TRIAL: NCT03412032
Title: Comparison of Two Summative Assessment Methods in Advanced Life Support Courses - a Randomized Controlled Trial
Brief Title: Comparison of Two Summative Assessment Methods in Advanced Life Support Courses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ILS_2017/2018
Record Dates: First submitted 2017-12-11; First posted 2018-01-26 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Self-Assessment
MeSH Terms: interventions — Restraint, Physical

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ERC (Other): Assessment as used by the European Resuscitation Council
  Interventions: Other: assessment
- AHA (Other): Assessment as used by the American Heart Association
  Interventions: Other: assessment

INTERVENTIONS:
Other: assessment — different assessments in both arms

SUMMARY:
Several approaches for summative assessment during Advanced Life Support courses are used. The most commonly used method during European Resuscitation (ERC) Council Life Support Courses is that 1 instructor is miming a whole team, and the candidate has to lead this "team" through a scenario; another variant of the summative assessment (mainly used by American Heart Association (AHA) Courses) is with a group of students, where one student is the team leader to be assessed and the others are his team not being assessed. The second approach might be more realistic; however there is no evidence around with regard to effectiveness (pass/fail rate, ability to test non-technical skills (NTS)) or participant/assessor satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* All medical students at the University of Bern, study year 2017/2018, 5th and 6th study year

Exclusion Criteria:

* Refusal to participate

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 428 (Actual)
Dates: Start 2017-12-02 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Team leadership | 1 minute after the assessment is completed
  Subjective rating of team leadership

CONTACTS AND LOCATIONS:
Overall Officials: Robert Greif, Study Chair — University of Bern, Switzerland
Locations (1):
- University of Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No